CLINICAL TRIAL: NCT01597531
Title: LIRAGLUTIDE AND ORLISTAT TREATMENT FOR PERSISTENT TYPE 2 DIABETES AFTER GASTRIC BANDING: A PILOT STUDY
Brief Title: Combinatorial Therapy for Peristent Type 2 Diabetes After Gastric Banding
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulty recruiting patients
Sponsor: East Carolina University (Other)
Responsible Party: Principal Investigator, Moahad S Dar, Assistant Professor of Medicine, East Carolina University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ECDOI-D71
Record Dates: First submitted 2012-05-10; First posted 2012-05-14 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Type 2 Diabetes; Gastric Banding
Keywords: Liraglutide; Orlistat
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Liraglutide; Orlistat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Liraglutide only (Active Comparator)
  Interventions: Drug: Liraglutide
- Orlistat only (Active Comparator)
  Interventions: Drug: Orlistat
- Liraglutide + Orlistat (Active Comparator)
  Interventions: Drug: Liraglutide + Orlistat

INTERVENTIONS:
Drug: Liraglutide — Liraglutide will be started at 0.6 mg injected subcutaneously daily for 1 week and then increased as tolerated to 1.2 mg and then a 1.8 mg daily.
  Arms: Liraglutide only
Drug: Orlistat — Orlistat will be started initially at a dose of 60 mg taken with the evening meal. Additional doses will be added at breakfast or lunch every 1-2 weeks as tolerated. The patient will be advised to skip drug dosing if little or no fat is contained in the meal. Target dose will 60 mg three times a day and the patients will be advised to take a multivitamin 2 hours before or after Orlistat addition to ensure adequate nutrition.
  Arms: Orlistat only
Drug: Liraglutide + Orlistat — Liraglutide will be started at 0.6 mg injected subcutaneously daily for 1 week and then increased as tolerated to 1.2 mg and then a 1.8 mg daily. Patients not tolerating a higher dose will be allowed to remain on the lower dose as long they tolerate the lower. Following titration of Liraglutide to a maximum tolerated dose, Orlistat will be started initially at a dose of 60 mg taken with evening meal. Additional doses will be added at breakfast or lunch every 1-2 weeks as tolerated. The patient will be advised to skip drug dosing if little or no fat is contained in the meal. Target dose will 60 mg three times a day.
  Arms: Liraglutide + Orlistat

SUMMARY:
The purpose of this study is to determine whether addition of 1 or 2 medicines after gastric banding can improve remission of type 2 diabetes.

DETAILED DESCRIPTION:
Liraglutide and Orlistat improve glycemic control by increasing glucagon-like-peptide-1 (GLP-1) response and fat malabsorption, respectively but do not reverse type 2 diabetes. Roux-en-y gastric bypass (RYGB) surgery reverses type 2 diabetes 84% of the time while the less invasive, reversible laparoscopic adjustable gastric banding (LAGB) procedure reverses type 2 diabetes 48% of the time.

Decreased caloric intake occurs after RYGB and LAGB but increased post-prandial GLP-1 response and fat malabsorption only occur after RYGB. Since FDA-approved agents Liraglutide and Orlistat increase GLP-1 response and fat malabsorption, respectively, it is of significant clinical interest to determine if addition of Liraglutide and/or Orlistat can improve type 2 diabetes remission rates in the 52% of patients who have not achieved diabetes reversal after gastric banding.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be eligible if they meet the following criteria:

* male or female,
* age 25-70 years,
* BMI 26-65,
* type 2 diabetic,
* weight stable for 3 months,
* status post laparoscopic adjustable gastric banding (LAGB) for at least 1 year,
* hemoglobin a1c 7-10%;
* on any diabetic regimen including insulin except for thiazolidinedione use in the past 6 months.

Exclusion Criteria:

Subjects will be excluded if they meet any of the following criteria:

* prior history of pancreatitis,
* prior history of gastroparesis,
* glomerular filtration rate (GFR) < 50,
* history of thyroid cancer/multiple endocrine neoplasia/thyroid nodules/medullary thyroid cancer,
* history of cholelithiasis,
* history of hyperoxaluria or calcium oxalate nephrolithiasis,
* abnormal AST,
* ALT elevation,
* current or past history of liver disease,
* history of Roux-en-y gastric bypass or gastric sleeve or any other bariatric procedure other than LAGB,
* type 1 diabetes,
* any gastrointestinal disease causing malabsorption (including but not limited to inflammatory bowel disease, celiac sprue),
* prior history of Orlistat or incretin therapy use in past 3 months,
* unwilling or unable to complete scheduled testing,
* thiazolidinedione use within past 6 months,
* any serious and/or unstable medical, psychiatric, or other condition(s) that prevents the patient from providing informed consent or complying with the study.

Patients who have had organ transplantation are on chronic anticoagulation, pregnant or have A1C values > 10% will also be excluded.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2012-06; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Type 2 diabetes remission | baseline, 1 and 4 months post-randomization
  Hemoglobin a1c will be used to assess type 2 diabetes remission.

SECONDARY OUTCOMES:
Whole body insulin sensitivity | baseline, 1 and 4 months post-randomization
  Minimal model testing will be used to assess whole body insulin sensitivity.
GLP-1 response | Baseline, 1 and 4 months post-randomization
  A mixed meal challenge will be used to assess meal-stimulated GLP-1 response.
First Phase Insulin secretion | Baseline, 1 and 4 months post-randomization
  Minimal model testing will be used to assess first phase insulin secretion.

CONTACTS AND LOCATIONS:
Locations (1):
- Brody School of Medicine at East Carolina University, Greenville, North Carolina, United States

REFERENCES:
- [Background] Buchwald H, Estok R, Fahrbach K, Banel D, Jensen MD, Pories WJ, Bantle JP, Sledge I. Weight and type 2 diabetes after bariatric surgery: systematic review and meta-analysis. Am J Med. 2009 Mar;122(3):248-256.e5. doi: 10.1016/j.amjmed.2008.09.041. PMID 19272486